CLINICAL TRIAL: NCT00905931
Title: Acute Oral Lycopene Therapy on Cerebral Autoregulation and Delayed Ischaemic Deficits Following Aneurysmal Subarachnoid Haemorrhage (LASH): A Randomized Controlled Trial
Brief Title: Lycopene Following Aneurysmal Subarachnoid Haemorrhage
Acronym: LASH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge Theranostics Ltd (Industry)
Responsible Party: Mr Peter John Kirkpatrick, Addenbrooke's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LASH 3
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Subarachnoid Hemorrhage; Aneurysm
Keywords: Aneurysmal subarachnoid hemorrhage (aSAH); Cerebral vasospasm; impaired cerebral autoregulation; transient hyperaemic response test; delayed ischaemic neurological deficits
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Vasospasm, Intracranial | interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Lycopene
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lycopene — 30 mg oral, daily, for 21 days
  Arms: Active
Drug: placebo — starch
  Arms: Placebo

SUMMARY:
In this study the investigators wish to explore the potential neuroprotective effects of acute oral supplementation of lycopene, a natural anti-oxidant derived from tomatoes, on cerebral vasospasm and autoregulation, and examine whether any improvements translate into a reduction of biochemical markers of vascular injury and inflammation a decrease in the prevalence of secondary strokes following subarachnoid haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years old,
* Confirmed aneurysmal subarachnoid hemorrhage (aSAH),
* Time from ictus < 96 hours

Exclusion Criteria:

* Age: < 18 years old,
* Non-aneurysmal SAH,
* Time from ictus > 96 hours,
* Severe carotid atherosclerotic disease (≥70%)
* High-dose statin therapy (>80 mg/day fluvastatin; >40 mg/day simvastatin; >40 mg/day pravastatin; >10 mg/day atorvastatin; >10 mg/day rosuvastatin 28),
* Allergy or hypersensitivity to tomatoes and tomato products and history of any other significant atopy/allergy (e.g. soy, whey, lutein, lecithin)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of vasospasm | Daily for 21 days
  Mean flow velocity in MCA > 120 cm/min; LR > 3 (4 if age < 50 years old)
Duration of impaired autoregulation measured with transcranial Doppler | Daily for 21 days
  Transient hyperaemic response test; Mx

SECONDARY OUTCOMES:
Level of biochemical markers of vascular injury: LDL, oxy-LDL, CRP, circulating endothelial cells, endothelial progenitor cells | Days: 0, 3, 6, 12, 14, 21

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Kirkpatrick, FRCS(SN), Principal Investigator — Division of Neurosurgery, Department of Clinical Neurosciences, University of Cambridge, Addenbrooke's Hospital, Hills Road, CB2 0QQ Cambridge, UK
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Verghese M, Sunkara R, Shackelford L, Walker LT. Lycopene and cardiovascular diseases. In Preedy VR, Watson RR Ed. Lycopene: nutritional, medicinal and therapeutic properties. Science Publishers, New Hampshire, USA 2008.